CLINICAL TRIAL: NCT00003686
Title: A Double Blind Phase III Study of Oral Pilocarpine for Opioid-Induced Dry Mouth
Brief Title: Pilocarpine in Treating Patients With Dry Mouth Caused by Opioids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to poor accrual.
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SC16; CAN-NCIC-SC16 (Other: PDQ); P-UPJOHN-CAN-NCIC-SC16 (Other: UPJOHN); CDR0000066788 (Other: PDQ unique registration number)
Record Dates: First submitted 1999-11-01; First posted 2004-08-17 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Oral Complications; Quality of Life
Keywords: oral complications; quality of life
MeSH Terms: interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilocarpine (Active Comparator)
  Interventions: Drug: pilocarpine hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pilocarpine hydrochloride — Pilocarpine 5 mg po qid x 4 weeks
  Arms: Pilocarpine
Drug: Placebo — Placebo 5 mg po qid x 4 weeks
  Arms: Placebo

SUMMARY:
RATIONALE: Pilocarpine may help to relieve dry mouth in patients receiving opioids for cancer therapy. It is not yet known whether pilocarpine is more effective than no further treatment for this condition.

PURPOSE: Randomized phase III trial to determine the effectiveness of pilocarpine in treating patients who have dry mouth caused by opioids.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effectiveness of daily oral pilocarpine versus placebo in relieving dry mouth due to the ongoing use of an opioid for cancer related pain at 2 weeks by comparing proportion of patients with at least one response during the 2 week period, time of first response, and duration of first response. II. Evaluate the adverse effects of pilocarpine in these patients. III. Evaluate whether constipation, sedation, poor appetite, and nausea are ameliorated by pilocarpine in these patients. IV. Evaluate the effect of pilocarpine on quality of life of this patient group. V. Determine the timing and duration of the effect of pilocarpine in this patient population.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients receive either oral pilocarpine four times daily (arm I) or oral placebo four times daily (arm II) for 4 weeks. At the end of the 4 weeks, all patients are given the option to receive oral pilocarpine. Quality of life is assessed 2 days prior to randomization, after 2 weeks of treatment, and after 4 weeks of treatment.

PROJECTED ACCRUAL: There will be 60 patients accrued into this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Complaint of dry mouth with ALL the following characteristics: At least 1 week in duration Attributed by the treating physician to an opioid Severity rating at least 20 mm on a 100 mm visual analog scale Must be receiving routine (i.e., not just as needed) dosing with one of the following opioids: morphine, hydromorphone, transdermal fentanyl, methadone, or oxycodone Intent to continue opioid therapy at the same or higher dose over the first 2 weeks that the patient is receiving protocol treatment

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-3 Life expectancy: At least 6 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Calcium less than 29.9 mg/dL Cardiovascular: No symptomatic congestive heart failure or hypotension (systolic blood pressure less than 100 mm Hg) Pulmonary: No obstructive pulmonary disease (asthma, chronic bronchitis, or chronic obstructive pulmonary disease) Other: No known sensitivity to pilocarpine No active oral candidiasis No Sjogren's syndrome No acute iritis or narrow-angle glaucoma Not pregnant or nursing Effective contraception required of all fertile patients Must be fluent and possess sufficient cognitive ability to complete quality of life questionnaires in either English or French without assistance from a caregiver

PRIOR CONCURRENT THERAPY: See Disease Characteristics Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to a field encompassing the parotid glands At least 1 week since prior radiotherapy to the chief site of pain No concurrent radiotherapy to chief site of pain for 2 weeks following randomization Surgery: Not specified Other: No concurrent tricyclic antidepressants (amitriptyline, nortriptyline, desipramine, or imipramine)

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1998-05-22 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy | 10 years
  To evaluate, using a 100 mm VAS, the effectiveness of oral pilocarpine 5 mg qid in relieving dry mouth due to the ongoing use of an opioid for cancer related pain at 2 weeks (day 15). This will include comparing the proportion of at least one response during the 2 week period, time to first response and duration of first response.

CONTACTS AND LOCATIONS:
Overall Officials: David Warr, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Humber River Regional Hospital, Weston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelhardt M, Dold SM, Ihorst G, Zober A, Moller M, Reinhardt H, Hieke S, Schumacher M, Wasch R. Geriatric assessment in multiple myeloma patients: validation of the International Myeloma Working Group (IMWG) score and comparison with other common comorbidity scores. Haematologica. 2016 Sep;101(9):1110-9. doi: 10.3324/haematol.2016.148189. Epub 2016 Jun 16. PMID 27479825